CLINICAL TRIAL: NCT00330525
Title: Pharmacodynamic Effects of Sibutramine on Gastric Function in Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1723-04
Record Dates: First submitted 2006-05-25; First posted 2006-05-29 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — sibutramine

INTERVENTIONS:
Drug: sibutramine

SUMMARY:
Control of food intake, size and frequency of meals are critical to the development of obesity. The stomach signals feelings of fullness after a meal and therefore plays a role in control of calorie intake. It is unclear whether the approved appetite reducing drug sibutramine changes the function of the stomach. Differences in the way individuals respond to treatment with the appetite suppressant sibutramine may also explain why some people lose weight while others do not.

This single center clinical study aims to compare functions of the stomach in healthy, overweight and obese individuals, and to evaluate the effects of the FDA-approved appetite suppressing medication sibutramine on weight loss and stomach functions in patients who are overweight or obese. The effect of individual differences in inherited genes on weight reduction with sibutramine will be tested.

DETAILED DESCRIPTION:
Background: Control of food intake, size and frequency of meals are critical to the development of obesity. The stomach signals satiation in response to calories and volume ingested, playing a role in control of calorie intake. It is unclear whether the approved appetite reducing drug sibutramine alters gastric physiology. Genetic variations are potentially key to inter-individual differences in responses to treatment with the appetite suppressant sibutramine.

Aims: 1. To compare gastric functions in healthy, overweight and obese individuals. 2. To evaluate effects of sibutramine on gastric functions and weight in patients who are overweight or obese. 3. To obtain preliminary data on the effect of genetic variation on responses to sibutramine.

Methods: We shall measure gastric emptying, fasting and postprandial gastric volumes (using validated, non-invasive imaging methods), postprandial satiation and satiety, and integrated plasma ghrelin, leptin, insulin, GLP-1 and peptide YY levels before and after 12 weeks of sibutramine 15mg vs. placebo. We shall also collect DNA, to eventually study effects of candidate genes on response to sibutramine.

Significance: Our study will provide the first evidence of the effects of sibutramine on gastric function.

ELIGIBILITY:
Inclusion Criteria

1. Normal weight, overweight and obese subjects with BMI> 18 Kg/m2 residing in Olmsted County, MN: Otherwise healthy individuals who are not currently on treatment for cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological, endocrine (other than hyperglycemia not requiring medical therapy) and unstable psychiatric disease.
2. Age: 18-65 years
3. Gender: Men or women. Women of childbearing potential will have negative pregnancy test within 48 h of enrollment and before each radiation exposure.

Exclusion Criteria

1. Weight exceeding 300 pounds or 137 kilograms (due to limitations regarding SPECT imaging studies).
2. Abdominal surgery other than appendectomy, Caesarian section or tubal ligation.
3. Positive history of chronic gastrointestinal diseases, systemic disease that could affect gastrointestinal motility or use of medications that may alter gastrointestinal motility, appetite or absorption e.g., orlistat (Xenical).
4. Significant psychiatric dysfunction based upon screening with the Hospital Anxiety and Depression Scale [HADS] self-administered alcoholism screening test (substance abuse) and the questionnaire on eating and weight patterns (binge eating disorders and bulimia). If such a dysfunction is identified by a HADS score >8 or difficulties with substance or eating disorders, the participant will be excluded and given a referral letter to his/her primary care doctor for further appraisal and follow-up.
5. Intake of medication, whether prescribed or OTC medication (except multivitamins) within 7 days of the study. Exceptions are birth control pill, estrogen replacement therapy, and thyroxine replacement.
6. Concomitant use of MAOI inhibitors and other centrally acting appetite suppressants (since this would make them ineligible for sibutramine treatment).
7. Hypersensitivity to sibutramine (since this would make them ineligible for sibutramine treatment).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2005-01; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
T1/2 gastric emptying of solids and liquids
Fasting whole gastric volume
Maximum volume of Ensure ingested (satiety testing)
weight loss in kg
effect of candidate SNPs/gene deletions on response to sibutramine

SECONDARY OUTCOMES:
Ghrelin, leptin, insulin, GLP-1, and PYY levels integrated over the 8 hours after the meal.
Aggregate symptom score 30 min after ingestion of Ensure
Body fat
Gastric residual at 2 and 4 hours; gastric emptying T10%, and parameters from power exponential analysis will also be described
Caloric intake from a standard ad libitum meal

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States